CLINICAL TRIAL: NCT04469647
Title: COVID 19 Antibody Seroprevalence Amongst Healthcare Workers in Johns Hopkins Aramco Healthcare
Brief Title: COVID 19 Seroprevalence Amongst Healthcare Workers in JHAH
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Johns Hopkins Aramco Healthcare (Other)
Responsible Party: Sponsor
Other Study IDs: IRB20-09
Record Dates: First submitted 2020-07-13; First posted 2020-07-14 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: COVID 19
Keywords: COVID 19; Coronavirus; SARS-CoV-2
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — Serologic Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- High-risk: Employees at high-risk of Coronavirus exposure areas (physicians, nurses, respiratory therapists, radiology technologists, lab technologists, housekeepers)
  Interventions: Diagnostic Test: Serology Test
- Low-risk: Employees working at lower risk areas such as (administration, HR, Public relations)
  Interventions: Diagnostic Test: Serology Test

INTERVENTIONS:
Diagnostic Test: Serology Test — Participants will be seen at T0 (baseline),T2 (2 months after T0), and T4 (2 months after T2).
  at every visit, participants will be asked to complete a general surveillance survey and a blood sample will be taken for the serology test.

SUMMARY:
Healthcare workers play a critical role in fighting the pandemic, not only by managing the patients' health clinically, but also by implementing adequate measures for infection prevention and control in healthcare facilities. This puts healthcare workers at a greater risk of acquiring the disease. COVID-19 is caused by Severe Acute Respiratory Syndrome Coronavirus -2 (SARS-CoV-2) and many people can be infected with it asymptomatically and undetectably.

Serology is an antibody test that provides additional information to polymerase chain-reaction (PCR) testing as it is the only way to reliably establish the fraction of the population that was infected . Seroconversion is the development of antibodies in the blood which can confirm suspected cases after the fact and reveal who was infected but asymptomatic and never realized it. Antibodies are specific proteins created as the body's response to the infection and this test is essential for detecting infected individuals with few or no symptoms at all.

ELIGIBILITY:
Inclusion Criteria:

1. Adult.
2. JHAH employee
3. Housekeepers (this group of staff are outsourced at JHAH)

Exclusion Criteria:

1. Any participant exhibiting COVID 19 symptoms

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthcare workers, divided into two groups (High-risk and Low-risk).
Sampling Method: Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2020-07-19 (Estimated); Primary Completion 2021-01-15 (Estimated); Study Completion 2021-06-15 (Estimated)

PRIMARY OUTCOMES:
Seroconversion status | 6 Months
  Percentage of health care workers with positive serological markers to describe patterns in exposure, re-infection, clinical symptom, serological responses among health care workers based on their baseline serological status over a one year period.

SECONDARY OUTCOMES:
The proportion of asymptomatic infections among staff who have seroconverted | 6 Months
  Seroconversion without clinical manifestation (fever, body aches, headache, sweating, chills + respiratory symptoms (cough dyspnea, sputum) or digestive (nausea / vomiting diarrhea abdominal pain)
The durability of COVID 19 seroconversion in asymptomatic healthcare workers at JHAH | 6 Months
  To identify the durability of antibody seroconversion
Identification of risk factors for COVID 19 seroconversion in asymptomatic healthcare workers | 6 Months
  Age, gender, type of staff, resources

CONTACTS AND LOCATIONS:
Locations (1):
- Johns Hopkins Aramco Healthcare, Dhahran, Eastern Province, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided
We are willing to share our data after collection de-identified. We plan to share the data with WHO for their unity studies

REFERENCES:
- [Derived] Mushcab H, Al-Tawfiq JA, Babgi A, Ghamdi M, Amir A, Sheikh SS, Darwisheh A, AlObaid A, Masuadi E, AlFattani A, Qahtani S, Al Sagheir A. Longevity of Immunoglobulin-G Antibody Response Against Nucleocapsid Protein Against SARS-CoV-2 Among Healthcare Workers. Infect Drug Resist. 2023 May 31;16:3407-3416. doi: 10.2147/IDR.S400365. eCollection 2023. PMID 37283943
- [Derived] Mushcab H, Al-Tawfiq JA, Ghamdi M, Babgi A, Amir A, Sheikh SS, Darwisheh A, Alobaid A, Jebakumar AZ, Qahtani S, Al Sagheir A. A Cohort Study of Seroprevalence of Antibodies Against SARS-CoV-2 Infection Among Healthcare Workers at a Tertiary Hospital in Saudi Arabia. Infect Drug Resist. 2022 Aug 10;15:4393-4406. doi: 10.2147/IDR.S369755. eCollection 2022. PMID 35974896
- See also: Coronavirus disease (COVID-19) technical guidance: The Unity Studies: Early Investigations Protocols — https://www.who.int/emergencies/diseases/novel-coronavirus-2019/technical-guidance/early-investigations